CLINICAL TRIAL: NCT05629000
Title: Cohort of Optimized Assessment Strategy of Carotid Artery Stenosis
Brief Title: Optimization Strategy of Carotid Artery Stenosis
Acronym: COAS-CAS
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUMCH-CAS-006
Record Dates: First submitted 2022-04-10; First posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-01

CONDITIONS: Carotid Artery Stenosis
Keywords: carotid artery stenosis; Perfusion; plaque; MRI; CT; PET/MRI; Ultrasound
MeSH Terms: conditions — Carotid Stenosis; Plaque, Amyloid | interventions — Endarterectomy, Carotid; Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plaques
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Carotid artery stenosis: patient with carotid artery stenosis
  Interventions: Procedure: Carotid revascularization; Diagnostic Test: MRI-PWI; Diagnostic Test: CTA; Diagnostic Test: PET/MRI; Diagnostic Test: Ultrasound

INTERVENTIONS:
Procedure: Carotid revascularization — All patients received carotid revascularization surgery at Peking Union Medical College Hospital.
  Other Names: carotid endarterectomy and carotid artery stent
Diagnostic Test: MRI-PWI — Multi-modal MRI before and after surgery.
Diagnostic Test: CTA — CTA before and after surgery.
Diagnostic Test: PET/MRI — PET/MRI before surgery.
Diagnostic Test: Ultrasound — Ultrasound before and after surgery.

SUMMARY:
The goal of this observational study is to learn about how to utilize multiple evaluation techniques in carotid artery stenosis patients for optimizing assessment of diagnosis and treatment strategy.

The main questions it aims to answer are:

* Identify best strategy that use multi-modal MRI and CT to assess patients' cerebral lesions and perfusion.
* Identify best strategy that use multi-modal MRI, PET-MRI ultrasound and CT to assess components and characters of patients' carotid plaques.

Participants will accept imaging examination before and after surgery. And doctors will collect basic characteristics, imaging results and biological samples of patients for analysis.

ELIGIBILITY:
Inclusion Criteria:

1. patients with severe stenosis (≥50%) or near-occlusion diagnosed by computed tomographic angiogram;
2. patients received carotid endarterectomy at Peking Union Medical College Hospital

Exclusion Criteria:

(1) Any contraindication to image examination; (3) refuse to sign the Informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Mild to severe carotid stenosis or near-occlusion patients receiving carotid revascularization treatment.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
stroke | During hospital stay, usually 7-30 days post operation
  perioperative stroke
cardiac infarction | During hospital stay, usually 7-30 days post operation
  perioperative cardiac infarction
transient ischemic attack | During hospital stay, usually 7-30 days post operation
  perioperative transient ischemic attack
cerebral hyperperfusion syndrome | During hospital stay, usually 7-30 days post operation
  perioperative cerebral hyperperfusion syndrome
death | During hospital stay, usually 7-30 days post operation
  perioperative death

SECONDARY OUTCOMES:
Image characters of MRI | half year after operation
  Arterial transit times, cerebral blood flow, plaque characters, etc.
Image characters of PET/MRI | half year after operation
  Diagnostic performance of 68Ga-FAPI PET/MR for intracranial or carotid atherosclerosis
Image characters of ultrasound | half year after operation
  Diagnostic performance of carotid artery ultrasound for intracranial or carotid atherosclerosis
Carotid plaque characters | half year after operation
  pathology characters of carotid plaque

CONTACTS AND LOCATIONS:
Locations (1):
- vascular surgery department of PUMCH, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lai Z, Wang C, Liu X, Sun H, Guo Z, Shao J, Li K, Chen J, Wang J, Lei X, Shu K, Feng Y, Kong D, Sun W, Liu B. Characterization of the proteome of stable and unstable carotid atherosclerotic plaques using data-independent acquisition mass spectrometry. J Transl Med. 2024 Mar 7;22(1):247. doi: 10.1186/s12967-023-04723-1. PMID 38454421